CLINICAL TRIAL: NCT05401747
Title: CONCERT STUDY: A Comprehensive ONline Program for Cognitive Enhancement, Reassurance and Training
Brief Title: A Comprehensive ONline Program for Cognitive Enhancement, Reassurance and Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 120314
Record Dates: First submitted 2022-05-10; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-04

CONDITIONS: Cognition Disorders in Old Age; Lifestyle, Healthy; Diet, Healthy; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy lifestyle intervention (Other): All cases will be assessed before and after intervention for cognitive changes.
  Interventions: Other: Healthy lifestyle

INTERVENTIONS:
Other: Healthy lifestyle — Nutrition consultation and teaching: A registered dietitian has the responsibility of teaching and explaining the diet. Plan: One meeting per 12 weeks. The exercise program is based on the Physical Activity Guidelines Advisory Committee and American Heart Association guideline and a modified version of Dose-Responses to Exercise Training study protocol for older adults summarized our weekly plans in detail. Plan: 2 meetings per week. Cognitive enhancement: Participants can select any of the following activities:methods requiring mental activities, physical activity, and social activity, enjoying music and our weekly dance classes (Waltz).

SUMMARY:
The CONCERT Study (A Comprehensive Online program for Cognitive Enhancement, Reassurance and Training) was designed to introduce a user-friendly platform to assess and train cognition among old adults.

Our main research questions are: i) Is it possible to provide a user-friendly platform to perform multi-domain cognitive training for old adults? ii) Are there any safety issues with these platforms? Inclusion criteria include: i) Aged ≥ 65 years; ii) Owning a computer with access to the Internet and basic knowledge to use it; iii) Having sufficient English language skill; iv) Normal baseline AD8 screening test; v) agree to join the study with their partners/ close family members.

Exclusion criteria include: i) History of dementia; ii) Severe physical disability precluding to participate in meetings; those using wheelchairs can still join the study with some modification in the exercise program.

Study duration includes 24 weeks of intervention with lifestyle changes (Online: Nutrition consultation and teaching, Exercise, dance, music therapy and cognitive enhancement). Participants have options to continue the study for another 24 weeks.

Outcome will be assessed based on participants' adherence, satisfaction.

DETAILED DESCRIPTION:
The CONCERT study is designed to provide an online platform for the public to provide healthy lifestyle recommendations and assess cognition. 60 participants (30 cases and 30 study partners) will be invited to this project. At baseline, all cases will be assessed with regard to cognition (AD8 Dementia Screening Interview), depression (Geriatric Depression Scale) and gait (Timed Up and Go). Participants will be asked to check their blood pressure at baseline and then every 3 months according to the Hypertension Canada's 2020 Guideline. All cases will be asked to participate in different educational classes, including nutrition consultation and teaching, exercise, dance (waltz), and music for 24 weeks. They will be also advised to accept the responsibility of a plant (Pothos, Spider Plant, Crocodile Fern and Aglaonema) at home. All meetings/ assessments are online. The investigators will assess adherence and satisfaction in all cases after 24 weeks. All cases will be invited to participate in another 24 weeks of intervention as an optional part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years;
* Owning a computer with access to the Internet and basic knowledge to use it;
* Having sufficient English language skill;
* Normal baseline AD8 screening test;
* Agree to join the study with their partners/ close family members. Age of family member or friend is not an exclusion criteria.

Exclusion Criteria:

* History of dementia;
* Severe physical disability precluding to participate in meetings; those using wheelchairs can still join the study with some modification in the exercise program;
* Active coronary heart disease or limitation for exercise based on their previous consults with their family physician/ cardiologists.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of online classes for healthy lifestyle. | 24 weeks and 50 weeks (optional) after initiation of the study
  To assess the adherence to online educational classes, each participant will receive a numeric code without any identifiers to join the meeting. The number of participants present in the meeting will be recorded to check for adherence. A booklet will be provided to the participants to note the programs used and their frequency during the week. The adherence to this study will be assessed using the trend test and Generalized Estimating Equation.

SECONDARY OUTCOMES:
Satisfaction of online classes for healthy lifestyle. | 24 weeks and 50 weeks (optional) after initiation of the study
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) will be used to evaluate participants' satisfaction. Patient's interest to participate in the second phase of the study (optional) and willingness to introduce the study to friends/ family members will be used as markers of total satisfaction.

IPD SHARING:
Plan to Share IPD: No
Data can be shared only after the Ethics approval.